CLINICAL TRIAL: NCT00419588
Title: Growth of Airways and Lung Parenchyma
Brief Title: Growth of Airways and Lung Tissues in Premature and Healthy Infants
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Robert Tepper, Robert Tepper, Indiana University
Other Study IDs: HL054062-09A1; 0512-20
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Infant, Premature, Diseases; Bronchopulmonary Dysplasia; Asthma
Keywords: infant, premature; Bronchopulmonary dysplasia; asthma
MeSH Terms: conditions — Infant, Premature, Diseases; Bronchopulmonary Dysplasia; Asthma; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal Cells are being obtained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1-Healthy Infants: Group 1: We have recruited 50 healthy infants born >37 weeks gestation, and between 2 and 36 months of age. Infants were excluded for any of the following reasons.
  1. Congenital cardio-respiratory disease
  2. Hospitalization for respiratory illness
  3. Treatment with asthma medications for more than one time
  4. Small for gestational age at birth
  5. More than one respiratory illness
  6. More than one episode of wheezing
- 3-Premature Infants: Group 3: We will recruit 115 infants born prematurely, 23-35 weeks gestation. Subjects will be evaluated at the corrected age between 2 and 24 months. The subjects will have no oxygen requirements, and be clinically stable outpatients when evaluated. Infants will be excluded for any of the following reasons.
  1. Congenital cardio-respiratory disease
  2. Severe developmental delay
- 2-Healthy Infants CT: Group 2: The investigators recruited 50 infants born at > 37 weeks gestation and they were evaluated between 2 and 36 months of age when scheduled for high resolution computed tomography (HRCT) imaging for non-respiratory medical problems. Subjects were enrolled and HRCT of the chest were obtained. Infants were excluded for the following reasons:
  1. Congenital cardio-respiratory disease
  2. Hospitalization for respiratory illness
  3. Treatment with asthma medications

SUMMARY:
The purpose of this study is to evaluate the growth of the lung and how easily gas can be taken up by the lung in healthy infants born at full term without any breathing problems and infants born prematurely.

DETAILED DESCRIPTION:
SPECIFIC AIM # 1: Determine the relationship between parenchymal tissue and alveolar volume with normal lung growth early in life We hypothesize that during the first two years of life that parenchymal surface area and alveolar volume increase with somatic growth; however, the ratio of surface area to volume remains constant, while ventilation within the lung becomes more homogenous.

SPECIFIC AIM # 2: Determine the pulmonary sequelae of premature birth and assess the effectiveness of early treatment strategies upon the pulmonary sequelae.

We hypothesize that premature birth impedes growth and development of the lung parenchyma and the airways at a corrected-age of 1-year. In addition, initiating continuous positive airway pressure (CPAP) and a permissive ventilatory strategy in very premature infants at birth will improve lung growth and lung function compared to treatment with early surfactant and conventional ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Group 1
* full term greater than 37 weeks
* Group 3
* infants born premature between 23-35 weeks of age to be tested between the ages of two to twenty four months corrected.

Exclusion Criteria:

* heart disease
* severe developmental delays

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: We are recruiting premature infants from Riley Hospial for Children, Methodist Hospital and IU NICu's. We also recruit from the Infant Lung Disease clinic at Riley Hospital for Children. Healhy full term infant are recruited through advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2006-09; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary function Test | day of testing
  Forced Expiratory flows, single breath diffusion capacity and alveolar volume

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Tepper, MD, PhD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States